CLINICAL TRIAL: NCT06028308
Title: The Effect of Adding Auditory Information on Head Movements in People With Traumatic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Associate Professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AAU031-1025976b
Record Dates: First submitted 2023-08-22; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Whiplash; Healthy
Keywords: Whiplash; Neck pain; Kinematics
MeSH Terms: conditions — Whiplash Injuries; Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sound 1 (Experimental): A sound will be played while moving the head
  Interventions: Device: Smartphone playing a sound
- Sound 2 (Experimental): A sound (different from Sound 1) will be played while moving the head
  Interventions: Device: Smartphone playing a sound
- No Sound (No Intervention): No sound will be played while moving the head

INTERVENTIONS:
Device: Smartphone playing a sound — A sound will be played from a portable device (smartphone mounted with earphones) during movement
  Arms: Sound 1; Sound 2

SUMMARY:
This study sets out to investigate the potential effect of auditory disturbances on human movement

DETAILED DESCRIPTION:
Clinicians routinely investigate/test human movement but if/how this is effect by auditory disturbances is unclear. This study sets out to investigate the impact of auditory disturbances on head movements.

ELIGIBILITY:
Control group:

Inclusion Criteria (Control):

* Able to speak, read and understand Danish/English

Exclusion Criteria (Control):

* Pain from the neck or shoulder area during the past 6 months
* Experience of delayed onset muscle soreness (DOMS) during the week leading up to the test session
* Former surgery in neck or shoulder
* Current or previous chronic or recurrent pain condition that could affect the results
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses that could affect the results
* Regular use of analgesics
* Abnormally disrupted sleep in the last 24 hours preceding the experiment
* Lack of ability to cooperate

Neck pain group:

Inclusion Criteria (Neck Pain):

* Traumatic onset of neck pain
* Able to speak, read and understand Danish/English
* Reduced/painful active range of motion of the head and/or painful reaction to palpation of the neck at the time of inclusion

Exclusion Criteria (Neck Pain):

* Experience of DOMS during the week leading up to the test session
* Former surgery in neck or shoulder
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal (other than neck pain) or mental illnesses that could affect the results
* Abnormally disrupted sleep in the 24 hours preceding the experiment
* Lack of ability to cooperate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | During a single test session (approximately 45minutes) at day 1
  Range of motion will be assessed during head rotations (i.e. moving the head from a neutral position to end of range in rotation before returning to the start position)

SECONDARY OUTCOMES:
Head repositioning accuracy | During a single test session (approximately 45minutes) at day 1
  Head repositioning accuracy will be assessed as the error between the starting point and the end point following a head rotation (i.e. moving the head from a neutral position to end of range in rotation before returning to the start position) and will be repressed in degrees.
Quality of head movement | During a single test session (approximately 45minutes) at day 1
  Quality of movement (smoothness) will be determined using calculations of jerk variance (Jerk is the time derivative of acceleration which will be measures using an inertial measurement unit. The measure will be converted to a unitless measure where higher values indicates less smooth movements), assessed during head rotations (i.e. moving the head from a neutral position to end of range in rotation before returning to the start position).
Perceived stiffness during movement | During a single test session (approximately 45minutes) at day 1
  Participants will rate their perceived stiffness during head movement using a 0-100 numerical rating scale, where 0 = no stiffness and 100 = worst stiffness imaginable.
Perceived difficultness of performing movement | During a single test session (approximately 45minutes) at day 1
  Participants will rate the Perceived difficultness of performing head movements using a 6-point Likert scale going from 0 = no problems, 1 = minimally difficult; 2 = somewhat difficult; 3 = fairly difficult; 4 = very difficult; 5 = unable to perform
Perceived neck pain intensity | During a single test session (approximately 45minutes) at day 1
  Participants will rate ant potential pain during the session using a 0-11 numeric rating scale (NRS) with 0 = no pain and 10 = worst imaginable pain

OTHER OUTCOMES:
Neck Disability Index (NDI) | At the beginning of the single test session (approximately 45minutes) at day 1
  The NDI questionnaire consists of 10 items (Domains: pain intensity, personal care, lifting, reading, headache, concentration, work, driving, sleeping, recreation) used to assess how neck pain affects your ability to manage everyday activities. Each item is score on a scale from 0-5 with a higher total score = high level of disability
Tampa Scale for Kinesiophobia (TSK-11) | At the beginning of the single test session (approximately 45minutes) at day 1
  The TSK-11 questionnaire consists of 11 items which is answered using a 4-point scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Score can range from 11 to 44 and a higher score indicated a greater kinesiophobia
Perceived area of neck pain | At the beginning of the single test session (approximately 45minutes) at day 1
  Participants will draw the area of perceived neck pain on a body chart
Fear Avoidance Beliefs Questionnaire-physical activity subscale (FABQpa) | Time Frame: At the beginning of the single test session (approximately 45minutes) at day 1
  The FABQpa subscale consists of 4 items which are used to assess the participants beliefs on how physical activity can affect their pain. The items are scored on a 7-point scale with 0 = Completely disagree and 6 = Completely agree. Score ranges from 0-24 with a higher score indicating higher fear avoidance beliefs with regards to physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Steffan WM Christensen, PhD, Principal Investigator — Aalborg University
Locations (2):
- Denmark (2):
  - FysioDanmark Aalborg, Aalborg
  - Dept. Of Health Science and Technology, Aalborg University, Gistrup